CLINICAL TRIAL: NCT04558476
Title: A Multicenter Randomized Trial to Assess the Efficacy of CONvalescent Plasma Therapy in Patients With Invasive COVID-19 and Acute Respiratory Failure Treated With Mechanical Ventilation: the CONFIDENT Trial
Brief Title: Efficacy of CONvalescent Plasma in Patients With COVID-19 Treated With Mechanical Ventilation
Acronym: CONFIDENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: KCE Belgian Healthcare Knowledge Centre (Unknown)
Responsible Party: Principal Investigator, Misset Benoit, Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003102-31
Record Dates: First submitted 2020-09-14; First posted 2020-09-22 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Covid19; Mechanical Ventilation Complication; Corona Virus Infection; Respiratory Failure; SARS (Severe Acute Respiratory Syndrome)
Keywords: Covid 19; Convalescent plasmatherapy; SARS Cov-2 pneumonia
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Insufficiency; Severe Acute Respiratory Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (Experimental): 2 units of plasma ( 400-500ml) from 2 different donnors duration of treatment =2 h
  Interventions: Biological: Convalescent Plasma
- Standard of care (Other): Standard of care according the last gold standards
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: Convalescent Plasma — 2 units of convalescent plasma
  Arms: Convalescent Plasma
Other: Standard of Care — Gold Standards
  Arms: Standard of care

SUMMARY:
The principal objective of the CONFIDENT trial is to assess the efficacy of two units (400-500 mL in total) of convalescent plasma, as compared to Standard of Care (SoC), to reduce day-28 mortality in patients with SARS-CoV-2 pneumonia who require mechanical ventilation.

DETAILED DESCRIPTION:
Design : multicenter randomized openlabel, phase II trial.

Number of patients to include : 500 (250 with plasma, 250 without plasma).

The principal objective is to assess the efficacy of the treatment to reduce day-28 mortality in patients with SARS-CoV-2 pneumonia who require mechanical ventilation.

Hypothesis: Passive immunization with plasma collected from patients having contracted COVID-19 and developed specific antibodies may alleviate symptoms and viral load of SARS-CoV-2 and reduce mortality.

The patients will receive currently accepted standard of care for both COVID-19 and usual organ dysfunctions observed in such cases. half the patients will be administered either Convalescent plasma, depending on the randomization process. All patients will be followed-up for one year after inclusion. The study will be considered either positive or negative, based on the principal objective. This means that the product convalescent plasme will be considered effective if mortality at day 28 is lower is patients treated with convalescent plasma than without it. The follow-up will allow to assess a series of secondary objectives, addressing the evolution of organ failures, viral infection, inflammatory response and long-term physical of psychological impact of COVID-19. Interim analyses will be performed every 100 patients included in order to stop the trial if an exceptionally good or bad result is observed, to prevent using or not using the product appropriately in further patients. These analyses will be supervised by an independent committee.

The choice to include only those patients under mechanical ventilation for severe respiratory failure makes this study different from other trials testing convalescent plasma, as most trial include less severe patients.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* hospitalization in an intensive care unit participating to the study
* medical diagnosis with SARS-CoV-2 pneumonia as defined by both:

  * extended interstitial pneumonia on CT scan or a chest X-ray, consistent with viral pneumonia, within 10 days prior to inclusion
  * Positive result of SARS-CoV-2 PCR test, or any emerging and validated diagnostic laboratory test for COVID-19, within 15 days prior to inclusion
* under mechanical ventilation administered through an endotracheal tube, for less than 5 days
* prior Clinical Frailty Scale < 6.
* written consent of the patient, or - if impossible - of a relative acting as the legal representative, or - if impossible - of a physician from a non-participating department of the same hospital acting as an impartial witness .

Exclusion Criteria:

* Pregnancy
* Prior episode of transfusion-related side effect
* Medical decision to limit therapy
* Current participation in another trial testing a COVID-19 therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Vital status | at day 28
  dead or alive

SECONDARY OUTCOMES:
day 90 mortality | at day 90
  dead or alive
number of ventilator-free days at day 28 | at day 28
  to assess the ventilator free days
number of renal replacement therapy free days at day 28 | at day 28
  to assess the number of renal replacement therapy free days
number of vasopressors free-days at day 28 | at day 28
  to assess the number of vasopressors free-days
use of ECMO before day 28 | till day 28
  to assess if ECMO was required
value of the SOFA score at days 7, 14 and 28 | Day 1, 7, 14, 28
  to assess the value of SOFA score
changes in SOFA scores (delta SOFA) over 7, 14 and 28 days | Day 7, 14 and 28 days
  to assess the changes in SOFA scores (delta SOFA)
assessment of the SARS-CoV-2 viral load | Days 7, 14 and 28
  assessment of the SARS-CoV-2 viral load, expressed as cycle threshold, [2] in the tracheal aspirates (for intubated patients) or nasopharyngeal swabs (for extubated patients) at days 7, 14 and 28
blood C reactive protein (CRP) concentration | Days 7, 14 and 28
  to assess the concentrations of C reactive protein (CRP)
ferritin concentration | Days 7, 14 and 28
  to assess the concentration of ferritin
lymphocyte count | Days 7, 14 and 28
  to assess the count of lymphocyte
length of stay in the acute care hospital | through study completion, 1 year
  to assess the lenght of stay in the acute care
location of the patient | Day 90
  to assess the location of the patient : acute care hospital, post acute care hospital, long-term residency, home
Katz Index of independence in Activity Day Living functional score | Day 90 and 365
  to assess the Activity Day Living functional Min value: 0 = Low (patient very dependent) Max value: 6 = High (patient independent)
Hospital Anxiety and Depression Scale (HADS) | Day 90 and 365
  to evaluate the anxiety-depression For each item 0-7 : Normal 8-10 : Bordeline abnormal (borderline case) 11-21 : Abnormal case
Quality of life scale EQ-5D-5L | Day 90 and 365
  The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.
Transfusion related adverse events | till 28 days
  to assess the transfusion related adverse events
Determine the type of concommittent inflammatory response | till 28 days
  assess clusters based on the profile of cytokines, chemokines and cell adhesion markers

CONTACTS AND LOCATIONS:
Locations (17):
- Belgium (17):
  - Clinique Saint Pierre Ottignies, Ottignies, Brabant Wallon
  - Centre Hospitalier Wallonie Picarde, Tournai, Hainaut
  - OLVZ Aalst, Aalst
  - UZ Antwerpen, Antwerp
  - Imelda ZH Bonheiden, Bonheiden
  - CHU Saint Pierre, Brussels
  - Erasme, Brussels
  - UZ Brussel, Brussels
  - CHU Charleroi Marie Curie, Charleroi
  - AZ Sint Blasius, Dendermonde
  - UZ Gent, Ghent
  - AZ Groeningen Kortrijck, Kortrijk
  - UC Louvain, Leuven
  - CHR Citadelle, Liège
  - CHU Liège, Liège
  - AZ Delta, Roeselare
  - CHU UCL Namur-Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Misset B, Diep AN, Bertrand A, Piagnerelli M, Hoste E, Michaux I, De Waele E, Dumoulin A, Jorens PG, van der Hauwaert E, Vallot F, Swinnen W, De Schryver N, de Mey N, Layios N, Mesland JB, Robinet S, Cavalier E, Donneau AF, Moutschen M, Laterre PF. Immunological sub-phenotypes and response to convalescent plasma in COVID-19 induced ARDS: a secondary analysis of the CONFIDENT trial. Ann Intensive Care. 2024 Oct 21;14(1):160. doi: 10.1186/s13613-024-01392-1. PMID 39432177
- [Derived] Misset B, Piagnerelli M, Hoste E, Dardenne N, Grimaldi D, Michaux I, De Waele E, Dumoulin A, Jorens PG, van der Hauwaert E, Vallot F, Lamote S, Swinnen W, De Schryver N, Fraipont V, de Mey N, Dauby N, Layios N, Mesland JB, Meyfroidt G, Moutschen M, Compernolle V, Gothot A, Desmecht D, Taveira da Silva Pereira MI, Garigliany M, Najdovski T, Bertrand A, Donneau AF, Laterre PF. Convalescent Plasma for Covid-19-Induced ARDS in Mechanically Ventilated Patients. N Engl J Med. 2023 Oct 26;389(17):1590-1600. doi: 10.1056/NEJMoa2209502. Epub 2023 Oct 25. PMID 37889107
- [Derived] Misset B, Hoste E, Donneau AF, Grimaldi D, Meyfroidt G, Moutschen M, Compernolle V, Gothot A, Desmecht D, Garigliany M, Najdovski T, Laterre PF. A multicenter randomized trial to assess the efficacy of CONvalescent plasma therapy in patients with Invasive COVID-19 and acute respiratory failure treated with mechanical ventilation: the CONFIDENT trial protocol. BMC Pulm Med. 2020 Dec 7;20(1):317. doi: 10.1186/s12890-020-01361-x. PMID 33287790